CLINICAL TRIAL: NCT06540066
Title: A Multicenter, Open-label, Phase 1a/1b Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-B3227 as Monotherapy and in Combination With Tislelizumab in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of BGB-B3227 Alone and in Combination With Tislelizumab in Participants With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-B3227-101; 2024-514216-27-00 (EU CTIS Number); CTR20244018 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Cancer; Advanced Solid Tumor; Metastatic Cancer; Metastatic Solid Tumor
Keywords: BGB-B3227; tislelizumab; BGB-A317; advanced solid tumor; metastatic solid tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — tislelizumab; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1a Part A: Dose Escalation (BGB-B3227 Monotherapy) (Experimental): Sequential cohorts of increasing dose levels of BGB-B3227 will be evaluated as monotherapy.
  Interventions: Drug: BGB-B3227
- Phase 1a Part B: Dose Escalation (BGB-B3227 + tislelizumab) (Experimental): Sequential cohorts of increasing dose levels of BGB-B3227 will be evaluated in combination with tislelizumab.
  Interventions: Drug: BGB-B3227; Drug: Tislelizumab
- Phase 1b: Dose Expansion (Experimental): Sequential cohorts of increasing dose levels of BGB-B3227 will be evaluated in combination with tislelizumab and chemotherapy.
  Interventions: Drug: BGB-B3227; Drug: Tislelizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: BGB-B3227 — Administered intravenously.
Drug: Tislelizumab — Administered intravenously.
  Other Names: BGB-A317
  Arms: Phase 1a Part B: Dose Escalation (BGB-B3227 + tislelizumab); Phase 1b: Dose Expansion
Drug: Chemotherapy — Administered in accordance with relevant local guidelines and/or prescribing information.
  Arms: Phase 1b: Dose Expansion

SUMMARY:
This is a first-in-human (FIH), open-label, multicenter dose escalation and expansion study of BGB-B3227, a humanized immunoglobulin G1 (IgG1) antibody. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BGB-B3227 as a monotherapy or in combination with tislelizumab with or without chemotherapy in participants with selected advanced or metastatic solid tumors. The study will also identify recommended dose(s) for expansion (RDFE[s]) of BGB-B3227 administered alone and in combination with tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumors with a high prevalence of mucin-1 (MUC1) expression
* At least 1 measurable lesion per RECIST v1.1
* Stable Eastern Cooperative Oncology Group Performance Status of ≤ 1
* Adequate organ function
* Willing to use a highly effective method of birth control

Exclusion Criteria:

* History of prior ≥ Grade 3 Cytokine Release Syndrome (CRS)
* History of severe Infusion-Related Reactions (IRRs), allergic reactions, or hypersensitivity to any ingredients or components of the study treatments
* Infection requiring systemic (oral or intravenous) therapy ≤ 14 days before the first dose of study drug(s), or participants with symptomatic COVID-19 infection
* Active leptomeningeal disease or uncontrolled, untreated brain metastasis
* Active autoimmune disease or history of autoimmune disease(s) that may relapse

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
Phase 1a: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From first dose of the study drug(s) to 30 days after the last dose or 90 days after last dose of tislelizumab, approximately 9 months
  Number of participants with AEs and SAEs, including findings from physical examinations, laboratory assessments, and that meet protocol-defined dose-limiting toxicity (DLT) criteria or protocol-defined Adverse Event of Special Interest (AESI) criteria.
Phase 1a: Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) | Approximately 9 months
  MTD is defined as the highest dose evaluated for which estimated toxicity rate is the closest to the target toxicity rate. MAD is defined as the highest dose administered if MTD is not reached.
Phase 1a: Recommended Dose(s) for Expansion (RDFE[s]) of BGB-B3227 | Approximately 9 months
  RDFE of BGB-B3227 alone or in combination with tislelizumab will be determined based upon the MTD or MAD.
Phase 1b: Objective Response Rate (ORR) | From first dose of study drug(s) until progressive disease or new anticancer treatment; approximately 12 months
  ORR is defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR), as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase 1b: Recommended Phase 2 Dose (RP2D) of BGB-B3227 | Approximately 12 months
  RP2D established from Phase 1a for BGB-B3227 for administration in combination with tislelizumab and chemotherapy in selected tumor types.

SECONDARY OUTCOMES:
Phase 1a: ORR | From first dose of study drug(s) until progressive disease or new anticancer treatment; approximately 6 months
  ORR is defined as the percentage of participants with confirmed best overall response of CR or PR, as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Phase 1b: Progression-Free Survival (PFS) | From first dose of study drug(s) until progressive disease or new anticancer treatment; approximately 12 months
  PFS is defined as the time from the first dose of study treatment to the date of first documentation of disease progression or death, whichever occurs first, as assessed by the investigator per RECIST Version 1.1.
Phase 1b: Number of Participants with AEs and SAEs | From first dose of the study drug(s) to 30 days after the last dose, or 90 days after last dose of tislelizumab; approximately 12 months
  Number of participants with AEs and SAEs, including findings from physical examinations, laboratory assessments, and that meet protocol-defined dose-limiting toxicity (DLT) criteria or protocol-defined Adverse Event of Special Interest (AESI) criteria.
Phase 1a and 1b: Disease Control Rate (DCR) | From first dose of study treatment drug(s) until confirmed response or stable disease; approximately 6 months for Phase 1a and 12 months for Phase 1b
  DCR is defined as the percentage of participants who achieve confirmed CR, PR, or stable disease, as assessed by the investigator per RECIST Version 1.1.
Phase 1a and 1b: Duration of Response (DoR) | From confirmed response to disease progression or death; approximately 6 months for Phase 1a and 12 months for Phase 1b
  DoR is defined as the time from the first confirmed objective response to disease progression documented after treatment initiation or death, whichever occurs first, as assessed by the investigator per RECIST Version 1.1.
Phase 1a and 1b: Serum Concentrations of BGB-B3227 | From first dose of BGB-B3227 up to 30 days after last dose of BGB-B3227; approximately 6 months for Ph1a and 12 months for Ph1b
Phase 1a and 1b: Number of Participants with Antidrug Antibodies (ADAs) against BGB-B3227 | From first dose of BGB-B3227 up to 30 days after last dose of BGB-B3227; approximately 6 months for Phase 1a and 12 months for Phase 1b
Phase 1a: Area under the Curve (AUC) of BGB-B3227 | Approximately 4 months
Phase 1a: Maximum observed plasma concentration (Cmax) of BGB-B3227 | Approximately 4 months
Phase 1a: Time to reach maximum observed plasma concentration (Tmax) of BGB-B3227 | Approximately 4 months
Phase 1a: Trough concentration (Ctrough) of BGB-B3227 | Approximately 4 months
Phase 1a: Accumulation ratio of BGB-B3227 | Approximately 4 months
Phase 1a: Terminal half-life (t1/2) of BGB-B3227 | Approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (12):
- United States (5):
  - Usc Norris Comprehensive Cancer Center (Nccc), Los Angeles, California
  - Washington University in St Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Next Oncology, Austin, Texas
  - Md Anderson Cancer Center, Houston, Texas
- China (3):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
- Italy (4):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Istituto Europeo Di Oncologia, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Istituto Clinico Humanitas, Rozzano

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/